CLINICAL TRIAL: NCT00108732
Title: A Phase II Study of PROSTVAC-V (Vaccinia)/TRICOM and PROSTVAC-F (Fowlpox)/TRICOM With GM-CSF in Patients With PSA Progression After Local Therapy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03075; NCI-2012-03075 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E9802; E9802 (Other: Eastern Cooperative Oncology Group); E9802 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2005-04-18; First posted 2005-04-19 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Prostate Carcinoma; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; PROSTVAC; rV-Tricom; sargramostim; Colony-Stimulating Factors

ARMS (1):
- Treatment (vaccine therapy) (Experimental): Patients receive vaccinia-PSA-TRICOM vaccine SC on day 1 and sargramostim (GM-CSF) SC on days 1-4 during weeks 1-4. Beginning in week 5, patients receive fowlpox-PSA-TRICOM vaccine SC on day 1 and GM-CSF SC on days 1-4. Treatment with fowlpox-PSA-TRICOM vaccine and GM-CSF repeats every 4 weeks for 3 courses (weeks 5-16). Beginning in week 17, patients receive fowlpox-PSA-TRICOM vaccine and GM-CSF as above every 12 weeks in the absence of clinical or biochemical disease progression or unacceptable toxicity.
  Patients with biochemical or clinical disease progression receive androgen ablation therapy comprising oral bicalutamide once daily for 1 month and goserelin SC once every 4 weeks in addition to fowlpox-PSA-TRICOM vaccine and GM-CSF. Treatment continues in the absence of further clinical or biochemical disease progression.
  Interventions: Drug: Bicalutamide; Drug: Goserelin Acetate; Biological: Recombinant Fowlpox-PSA(L155)/TRICOM Vaccine; Biological: Recombinant Vaccinia-TRICOM Vaccine; Biological: Sargramostim

INTERVENTIONS:
Drug: Bicalutamide — Given orally
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Biological: Recombinant Fowlpox-PSA(L155)/TRICOM Vaccine — Given SC
  Other Names: PROSTVAC-F; rFowlpox-PSA(L155)/TRICOM Vaccine
Biological: Recombinant Vaccinia-TRICOM Vaccine — Given SC
  Other Names: rV-TRICOM; Vaccinia-TRICOM; vaccinia-TRICOM vaccine
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells. Biological therapies, such as GM-CSF, may stimulate the immune system in different ways and stop tumor cells from growing. Androgens can cause the growth of prostate cancer cells. Drugs, such as bicalutamide and goserelin, may stop the adrenal glands from making androgens in patients whose tumor cells continue to grow. Giving vaccine therapy together with GM-CSF and, when needed, androgen ablation may be a more effective treatment for prostate cancer. This phase II trial is studying how well giving vaccine therapy together with GM-CSF works in treating patients with prostate cancer that progressed after surgery and/or radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect of PROSTVAC-V/TRICOM (Vaccinia) on cycle 1 followed by PROSTVAC-F/TRICOM (Fowlpox) and GM-CSF on biochemical PSA progression at 6 months.

II. To determine the change in PSA velocity pre-treatment to post-treatment.

SECONDARY OBJECTIVES:

I. To evaluate the percentage of patients experiencing a >50% decline in serum PSA repeated at 4 weeks.

II. To evaluate tolerability and any toxicity related to treatment with PSA vaccine and GM-CSF.

III. To determine the effect of GM-CSF on PSA immediately after treatment (day 4) compared to a delayed effect (day 15).

IV. To determine the PSA nadir, and percentage of patients with undetectable PSA, treated with combined vaccine and androgen ablation therapy over 12 months.

OUTLINE: This is a multicenter study.

Patients receive vaccinia-PSA-TRICOM vaccine subcutaneously (SC) on day 1 and sargramostim (GM-CSF) SC on days 1-4 during weeks 1-4. Beginning in week 5, patients receive fowlpox-PSA-TRICOM vaccine SC on day 1 and GM-CSF SC on days 1-4. Treatment with fowlpox-PSA-TRICOM vaccine and GM-CSF repeats every 4 weeks for 3 courses (weeks 5-16). Beginning in week 17, patients receive fowlpox-PSA-TRICOM vaccine and GM-CSF as above every 12 weeks in the absence of clinical or biochemical disease progression or unacceptable toxicity.

Patients with biochemical or clinical disease progression receive androgen ablation therapy comprising oral bicalutamide once daily for 1 month and goserelin SC once every 4 weeks in addition to fowlpox-PSA-TRICOM vaccine and GM-CSF. Treatment continues in the absence of further clinical or biochemical disease progression.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 10 years.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven prostate cancer and tumors limited to the prostate (including seminal vesical involvement, provided all visible disease was surgically removed) that have completed local therapy and have an elevated PSA after surgery or rising PSA after radiation therapy, as defined below; patients with lymph node involvement (D1) are not eligible
* Histologically confirmed diagnosis of prostate cancer
* Previous treatment with definitive surgery or radiation therapy or both
* No evidence of metastatic disease on physical exam, CT (MRI), and bone scan within 4 weeks prior to randomization
* Prior neoadjuvant/adjuvant hormonal or chemotherapy is allowed if it was last used >= 1 year prior to enrollment (no prior vaccine/immunotherapy for prostate cancer will be allowed)
* No therapy modulating testosterone levels (such as leuteinizing-hormone releasing-hormone agonists/antagonists and antiandrogens) is permitted within 1 year prior to enrollment; agents such as 5-reductase inhibitors, ketoconazole, megestrol acetate, systemic steroids, and herbal products are not permitted at any time during the period that the PSA values are being collected
* Hormone-sensitive prostate cancer as evident by a serum total testosterone level > 150 ng/dL at the time of enrollment within 4 weeks prior to randomization
* There must be one PSA measurement (referred to as the baseline PSA) obtained within one week prior to registration; the baseline PSA value must be greater than 0.4 ng/mL (after prostatectomy) or greater than 1.5 ng/mL (after radiation therapy)
* All patients must have evidence of biochemical progression as determined by 3 PSA measurements (PSA1, PSA2, PSA3), each higher than the previous value, each obtained at least 4 weeks apart from the others with the most recent one (PSA3) being the baseline PSA; all of these PSA values must be obtained at the same reference lab; the earliest (PSA1) must be done within 6 months prior to registration.
* PSA doubling time (PSADT) must be less than 12 months, calculated using the following formula:

PSADT in days = (0.693 (t))/(In (PSA3) - In (PSA2)) Where t = the number of days between PSA3 and PSA2 In = the natural log PSADT in months = PSADT in days divided by 30.4375

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 1
* Leukocytes >= 3000/mm^³
* Granulocytes >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine within normal institutional limits or creatinine clearance >= 60 mL/min for patients with creatinine levels above institutional normal (a calculated clearance may be used); an initial urine analysis will be required with grade 0 proteinuria and no abnormal sediment; for any positive protein a 24 hour urine should be less than 1,000 mg per 24 hours and no indication of chronic renal disease
* Serum total bilirubin, and alkaline phosphatase within normal institutional limits
* SGOT (AST) and SGPT (ALT) =< 2.5 x institutional upper limit of normal
* Patients cannot have evidence of immunosuppression:

  * Patients must be human immunodeficiency virus sero-negative due to the potential for severe reactions to vaccinia and the need for an intact immune system to respond to the immunization
  * Patients must not have active autoimmune diseases such as Addison's disease, Hashimoto's thyroiditis, systemic lupus erythematous, Sjogren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome or active Grave's disease; patients with a history of autoimmunity that has required systemic immunosuppressive therapy or has impaired organ function including CNS, heart, lungs, kidneys, skin, and GI tract are ineligible; patients receiving replacement thyroid hormone would be eligible
  * No concurrent use of systemic steroids, except for local (topical, nasal, or inhaled) steroid use; steroid eye drops are contraindicated for at least 2 weeks before vaccinia vaccination and at least 4 weeks post vaccinia vaccination
  * Patients must be hepatitis B and hepatitis C negative
* Patients must have a normal PT/INR within 4 weeks prior to randomization
* Patients must not be receiving any other investigational agents or receiving concurrent anticancer therapy
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; because of the recently recognized risk of cardiac inflammation after vaccinia, patients with clinically significant cardiomyopathy are excluded; patients must have recovered from any intercurrent illness and any acute toxicity related to prior therapy (i.e., surgery and/or radiation)
* Patients must use a safe and effective method of contraception to prevent virus transmission; the potential risk to spermatogenesis and fetal development after paternal immunization with this vaccine is not known; patients must agree to avoid fathering a child and use a latex barrier with adequate contraception prior to study entry and for at least 4 months following the last vaccine injection
* All sites of disease must be evaluated within 4 weeks prior to registration
* Patients with significant allergy or hypersensitivity to eggs should be excluded; patients must not have a history of allergy or untoward reaction to prior vaccination with vaccinia virus or to any component of the vaccinia vaccine regimen
* Patients must not have active eczema, a history of eczema, atopic dermatitis, or Darier.s disease; other acute, chronic, or exfoliative skin conditions (e.g., burns, impetigo, varicella zoster, severe acne, contact dermatitis, psoriasis, herpes or other open rashes or wounds
* Patients must be able to avoid close contact with those who share housing or have close physical contact for at least three weeks after recombinant vaccinia vaccination with persons at increased risk including those with active or a history of eczema or atopic dermatitis, or Darier"s disease; those with other acute, chronic or exfoliative skin conditions (e.g., burns, impetigo, varicella zoster, severe acne, contact dermatitis, psoriasis, herpes or other open rashes or wounds) until condition resolves; pregnant or nursing women; children 3 years of age and under; and immunodeficient or immunosuppressed persons (by disease or therapy), which includes those infected with HIV until the condition resolves

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert DiPaola, Principal Investigator — Eastern Cooperative Oncology Group
Locations (7):
- United States (7):
  - Baptist Cancer Institute, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Eastern Cooperative Oncology Group, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University Langone Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on February 3, 2006 and terminated on December 11, 2007 after reaching its accrual goal. A total of 50 patients were recruited from ECOG member institutions.
  Patients with biochemical or clinical progression during Step 1 were eligible to receive androgen blockade in Step 2. To date, 31 patients have registered to Step 2.
Groups:
- Vaccinia/Fowlpox/GM-CSF: There are two steps in this study. Patients receive vaccine treatment in Step 1. Patients with biochemical or clinical progression during Step 1 were eligible to continue on to androgen blockade in Step 2. This report includes information collected in Step 1 only.
  Patients receive vaccinia subcutaneously (SC) on day 1 and GM-CSF SC on days 1-4 during cycle 1. Beginning with cycle 2, patients receive fowlpox SC on day 1 and GM-CSF SC on days 1-4. Treatment with fowlpox and GM-CSF repeats every 4 weeks for 2 courses. Beginning in week 13, patients receive fowlpox and GM-CSF as above every 12 weeks in the absence of clinical or biochemical disease progression or unacceptable toxicity.
  Patients with biochemical or clinical disease progression may start Step II androgen ablation therapy comprising oral bicalutamide once daily for 1 month and goserelin SC once every 4 weeks in addition to fowlpox vaccine and GM-CSF until further progression or a max of 12 months.
Period: Step 1 (Vaccinia/Fowlpox/GM-CSF)
Arm/Group | Vaccinia/Fowlpox/GM-CSF
Started | 50
Eligible and Treated | 40
Completed | 36
Not Completed | 14
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Ineligible | 10
Not completed — Non-compliance | 1
Period: Step 2 (Androgen Ablation and Vaccine)
Arm/Group | Vaccinia/Fowlpox/GM-CSF
Started | 31
Completed | 26
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Groups:
- Vaccinia/Fowlpox/GM-CSF: Patients receive vaccinia subcutaneously (SC) on day 1 and GM-CSF SC on days 1-4 during cycle 1. Beginning with cycle 2, patients receive fowlpox SC on day 1 and GM-CSF SC on days 1-4. Treatment with fowlpox and GM-CSF repeats every 4 weeks for 2 courses. Beginning in week 13, patients receive fowlpox and GM-CSF as above every 12 weeks in the absence of clinical or biochemical disease progression or unacceptable toxicity.
  Patients with biochemical or clinical disease progression may start androgen ablation therapy comprising oral bicalutamide once daily for 1 month and goserelin SC once every 4 weeks in addition to fowlpox vaccine and GM-CSF until further progression or a max of 12 months.
Arm/Group | Vaccinia/Fowlpox/GM-CSF
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 62.5 [48 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Free of PSA Progression at 6 Months (Prior to the Start of Androgen Ablation)
Description: For patients who achieved a > 50% decline in PSA, an increase in PSA value by 50% over the nadir, confirmed by a second PSA two weeks later is considered progressive disease. The PSA rise must be at least 5 ng/mL or back to pretreatment baseline, whichever is greater.
  Changes in PSA below 5 ng/mL will not be considered assessable for progression.
  For patients whose PSA has not decreased by 50%, an increase in PSA value > 50% of baseline (on trial) or nadir PSA, whichever is lower, confirmed by a repeat PSA two weeks later is considered progressive disease. The PSA must have risen by at least 5 ng/mL.
Time Frame: Assessed at 6 months
Population: Only eligible and treated patients in step I are included in this analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of patients
Arm/Group | Vaccinia/Fowlpox/GM-CSF
Number analyzed (Participants) | 40
Proportion of patients | 0.625 [0.483 to 0.753]
Statistical Analysis 1: Comparison: Vaccinia/Fowlpox/GM-CSF; Test type: Superiority or Other; Percent = 62.5, 90% CI 2-sided [48.3 to 75.3]

2. Secondary Outcome: Proportion of Patients With PSA Response
Description: PSA response is defined as complete biochemical response or partial response.
  Complete Response:
  A PSA < 0.2 ng/mL confirmed by a repeat PSA one month later is considered a complete biochemical response for patients with prior radical prostatectomy. A PSA < 1 ng/mL on three separate occasions taken at least one month apart is considered a complete biochemical response in patients with radiation therapy only.
  Partial Response:
  A reduction in PSA by > 50% from baseline, confirmed by repeat PSA 1 month later.
Time Frame: Assessed monthly during the first 24 weeks and then every 3 months for a maximum total of 24 months
Population: Only eligible and treated patients in step I are included in this analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of patients
Arm/Group | Vaccinia/Fowlpox/GM-CSF
Number analyzed (Participants) | 40
Proportion of patients | 0 [0.0 to 0.072]
Statistical Analysis 1: Comparison: Vaccinia/Fowlpox/GM-CSF; Test type: Superiority or Other; Response rate (percent) = 0, 90% CI 2-sided [0 to 7.2]

3. Secondary Outcome: Difference Between Day 4 PSA Level and Day 15 PSA Level
Description: PSA level was assessed on Day 4 and Day 15 of cycle 1, and a comparison between the two measurements was done.
Time Frame: Assessed at day 4 and day 15 of cycle 1
Population: Only 22 patients with both day 4 and day 15 PSA levels available were included in this analysis.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Vaccinia/Fowlpox/GM-CSF
Number analyzed (Participants) | 22
ng/mL | 0.45 [-1.7 to 2.4]
Statistical Analysis 1: Comparison: Vaccinia/Fowlpox/GM-CSF; Test type: Superiority or Other; p = 0.003, Wilcoxon signed rank test; The Wilcoxon signed rank test was used to test the difference between day 4 PSA and day 15 PSA; median of difference = 0.45

4. Secondary Outcome: The Difference Between PSA Slopes Before and After Treatment
Description: PSA slopes were assessed by multiple PSA values obtained prior to registration and during treatment. Only patients who completed at least 3 months of treatment were included in this analysis. The PSA slopes were calculated by a piecewise linear model using the three or four PSA values obtained prior to registration and PSA measurements obtained every 4 weeks for the first six months of treatment. Natural log transformed PSA levels were used in this analysis, and the difference between PSA slopes before and after treatment was calculated.
Time Frame: Assessed monthly during the first 24 weeks and then every 3 months for a maximum total of 24 months
Population: Only 31 patients who completed at least 3 months of treatment were included in this analysis.
Measure: Median (Full Range); unit: log PSA/month
Arm/Group | Vaccinia/Fowlpox/GM-CSF
Number analyzed (Participants) | 31
log PSA/month | -0.04 [-0.30 to 0.18]
Statistical Analysis 1: Comparison: Vaccinia/Fowlpox/GM-CSF; Test type: Superiority or Other; p = 0.02, Wilcoxon signed rank test — The Wilcoxon signed-rank test was used to test the difference between pre and post-treatment PSA slopes assessed by multiple PSA values on natural log scale using a piecewise linear model with a common knot point at the date of registration; median of difference = -0.04

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment.
Arm/Group | Vaccinia/Fowlpox/GM-CSF
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 44/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccinia/Fowlpox/GM-CSF (N=50)
Fever w/o neutropenia (General disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Muscle pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccinia/Fowlpox/GM-CSF (N=50)
Anemia (Blood and lymphatic system disorders) | 4
Fatigue (General disorders) | 20
Fever w/o neutropenia (General disorders) | 14
Rigors/chills (General disorders) | 7
Injection site reaction (General disorders) | 28
Hot flashes (Vascular disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Bilirubin increased (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 6
Joint pain (Musculoskeletal and connective tissue disorders) | 3
Muscle pain (Musculoskeletal and connective tissue disorders) | 21
Pain-other (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less